CLINICAL TRIAL: NCT05597774
Title: Effects of Respiratory Muscle Training Combined With an Exercise Training Program in Individuals With Long-term Post-COVID-19 Symptoms
Brief Title: Effects of Respiratory Muscle Training in Individuals With Long-term Post-COVID-19 Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Colegio Profesional de Fisioterapeutas de la Comunidad de Madrid (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21/747
Record Dates: First submitted 2022-10-07; First posted 2022-10-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2022-09

CONDITIONS: Covid19; Post-acute COVID-19 Syndrome
Keywords: Respiratory Muscle Training; Tele-rehabilitation; Quality of Life; Exercise
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome; Motor Activity | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training + Inspiratory and expiratory muscle training group (Experimental): Participants will perform a cardiovascular exercise program 2 days per week during 8 weeks in the hospital, combined with an inspiratory and expiratory muscle training by a threshold device at home, twice a day, 3 days per week, for 8 weeks supervised by a physiotherapist through a virtual platform.
  Interventions: Other: Inspiratory + expiratory muscle training group; Other: Exercise training program
- Exercise training + Inspiratory and expiratory muscle training sham group (Sham Comparator): Participants will perform a cardiovascular exercise program 2 days per week during 8 weeks in the hospital, combined with an inspiratory and expiratory muscle training by a sham threshold device at home, twice a day, 3 days per week, for 8 weeks supervised by a physiotherapist through a virtual platform.
  Interventions: Other: Inspiratory + expiratory muscle training sham group; Other: Exercise training program

INTERVENTIONS:
Other: Inspiratory + expiratory muscle training group — Participants will perform an inspiratory and expiratory muscle training including warm-up, recovery between intervals and return to calm.
  Arms: Exercise training + Inspiratory and expiratory muscle training group
Other: Inspiratory + expiratory muscle training sham group — Participants will perform an inspiratory and expiratory muscle training including warm-up, recovery between intervals and return to calm.
  Arms: Exercise training + Inspiratory and expiratory muscle training sham group
Other: Exercise training program — Participants will perform a cardiovascular exercise program including warm-up, recovery between intervals and return to calm by cycloergometer.

SUMMARY:
The main objective of the present study is to observe the short-term effects of respiratory muscle training combined with an exercise training program on quality of life and exercise tolerance in individuals with long-term post-COVID-19 symptoms. As secondary objectives, the effects on respiratory muscle function, physical and lung function, as well as on the psychological state of these individuals.

DETAILED DESCRIPTION:
It is a double-blind randomized clinical trial study. Each participant will be randomly assigned to one of the following groups: 1) Exercise training program + Inspiratory muscle training + Expiratory muscle training, 2) Exercise training program + Sham Inspiratory muscle training + Sham Expiratory muscle training.

The exercise training program will be delivered in hospital and will be applied 2 sessions per week during 8 weeks. The exercise component will be lasted for 1hour and it consisted of cardiovascular exercises.

The respiratory muscle training program will be applied twice a day, 3 sessions per week during 8 weeks by a threshold device. The evening sessions will be supervised by a physiotherapist through a virtual platform.

Participants received baseline assessments at the beginning of the intervention and post-intervention assessments at the end of the 8th week.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years who presented long-term post-COVID-19 symptoms of fatigue and dyspnoea for at least 3 months after the COVID-19 diagnosis

Exclusion Criteria:

* Progressive respiratory, neuromuscular or neurological disorders and/or psychiatric or cognitive conditions that hindered their ability to cooperate
* Comorbidity that could interfere with the study interventions
* Any contraindication to the training interventions
* Previous inclusion in a rehabilitation program for their long-term post-COVID-19 symptoms (previous 3 months)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Change in quality of life | Baseline and 1-week post-intervention (9 weeks from baseline)
  Change in quality of life between baseline and post-intervention, as measured by the EuroQol-5D questionnaire which consists of 5 dimensions with 5 response options based on severity level, ranging from 1 to 5. An index score is provided, ranging from 0 (death) to 1 (full health).
Change in exercise tolerance | Baseline and 1-week post-intervention (9 weeks from baseline)
  Change in exercise tolerance between baseline and post-intervention, as measured by a cardiopulmonary exercise test

SECONDARY OUTCOMES:
Change in respiratory muscle function | Baseline and 1-week post-intervention (9 weeks from baseline)
  Change in inspiratory/expiratory muscle strength and inspiratory muscle endurance between baseline and post-intervention, as measured by maximum static inspiratory and expiratory pressures and by a constant load breathing test
Change in physical function | Baseline and 1-week post-intervention (9 weeks from baseline)
  Change in lower and upper limb strength between baseline and post-intervention, as measured by 1-min Sit-to-Stand and peripheral muscle force (dynamometry)
Change in pulmonary function | Baseline and 1-week post-intervention (9 weeks from baseline)
  Change in pulmonary function and diffusion capacity for carbon monoxide between baseline and post-intervention, as measured by pulmonary function tests
Change in psychological status | Baseline and 1-week post-intervention (9 weeks from baseline)
  Change in anxiety/depression levels between baseline and post-intervention, as measured by Hospital Anxiety and Depression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Ibai López de Uralde, PhD, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Hospital Universitario 12 de Octubre de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McNarry MA, Berg RMG, Shelley J, Hudson J, Saynor ZL, Duckers J, Lewis K, Davies GA, Mackintosh KA. Inspiratory muscle training enhances recovery post-COVID-19: a randomised controlled trial. Eur Respir J. 2022 Oct 6;60(4):2103101. doi: 10.1183/13993003.03101-2021. Print 2022 Oct. PMID 35236727
- [Background] Nopp S, Moik F, Klok FA, Gattinger D, Petrovic M, Vonbank K, Koczulla AR, Ay C, Zwick RH. Outpatient Pulmonary Rehabilitation in Patients with Long COVID Improves Exercise Capacity, Functional Status, Dyspnea, Fatigue, and Quality of Life. Respiration. 2022;101(6):593-601. doi: 10.1159/000522118. Epub 2022 Feb 24. PMID 35203084
- [Derived] Del Corral T, Fabero-Garrido R, Plaza-Manzano G, Izquierdo-Garcia J, Lopez-Saez M, Garcia-Garcia R, Lopez-de-Uralde-Villanueva I. Effect of respiratory rehabilitation on quality of life in individuals with post-COVID-19 symptoms: A randomised controlled trial. Ann Phys Rehabil Med. 2025 Feb;68(1):101920. doi: 10.1016/j.rehab.2024.101920. Epub 2025 Jan 11. PMID 39798250